CLINICAL TRIAL: NCT03097419
Title: The Effect of Remote Ischemic Conditioning on the Metabolomic Profile of NSTEMI Patients
Brief Title: Ischemic Conditioning in STEMI Patients
Acronym: EDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Nathan Shapiro, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012P000095
Record Dates: First submitted 2015-09-08; First posted 2017-03-31 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Arrest
Keywords: non-ST segment elevation myocardial infarction; myocardial infarction; remote ischemic conditioning; ischemic conditioning; sphygmomanometer; metabolomics
MeSH Terms: conditions — Heart Arrest; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: We will perform a prospective, randomized-controlled study of 300 patients presenting to the BIDMC ED with a suspected non-ST segment elevation myocardial infarction. After obtaining consent, the patients will be assigned to either the intervention or standard of care group via a computerized block 1:1 randomization process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Remote post-ischemic conditioning
  Interventions: Procedure: Remote post-ischemic conditioning
- Control (No Intervention): Standard medical care by the primary treatment team.

INTERVENTIONS:
Procedure: Remote post-ischemic conditioning — A manual sphygmomanometer will be inflated over the brachial artery of the participants' arm that does not have an intravenous catheter actively infusing medications. If both arms are in use, then the participant's non-dominant arm will be used.
  * The sphygmomanometer will be inflated to a pressure at least 20 mmHg greater than the participants' last recorded systolic blood pressure.
  * The sphygmomanometer will be inflated for 5 minutes then rapidly deflated for 5 minutes, thereby concluding one iteration.
  * Five (5) total iterations constitute the treatment.
  * The left arm will be preferentially used instead of the right arm, unless the left arm is receiving medication administration.
  Arms: Intervention

SUMMARY:
The purposes of the study are to 1) study alterations in the metabolomic profile of patients exposed to post-ischemic conditions and 2) study alterations in myocardial infarction size of patients exposed to post-ischemic conditioning.

DETAILED DESCRIPTION:
Myocardial infarction is a common, morbid and mortal disease. This study will examine both the clinical effects of the treatment as well as the molecular mechanism. Evaluating patients in the emergency department (ED) is more than a daily occurrence for every practicing emergency physician in the country. Every year there are approximately 4.5 million visits to the ED for chest pain and over 1.5 million hospitalizations for acute coronary syndrome (ACS).2 Despite its prevalence, ACS is a difficult diagnosis to evaluate and manage; it involves taking a thorough history and performing a physical as well as performing an electrocardiogram (ECG) and biomarker analysis. The pathogenesis of unstable angina and non-ST segment elevation myocardial infarctions (NSTEMI) involves occlusive narrowing of a coronary artery, usually from an atherosclerotic plaque. The downstream effect of which is inadequate oxygen delivery to the myocardium, resulting in cell death.

Ischemic conditioning is the protective mechanism by which brief episodes of ischemia protect the heart from ischemia-reperfusion injury. There are two types of ischemic conditioning commonly referred to in the literature: pre-conditioning and post-conditioning. In the example of pre-operative coronary artery bypass graft (CABG) patients who may experience a degree of ischemia peri-operatively, ischemic conditioning can be performed before the surgery to prevent or limit myocardial injury. In the example of a patient with an ongoing STEMI who is going to the interventional cardiology suite for a percutaneous intervention, post-ischemic conditioning therapy may prevent or limit myocardial injury. A "remote" qualifier specifies that the therapy is implemented by inducing ischemia at a location that is not the heart itself.

The investigators propose to leverage the novel technique of metabolomics to better study the mechanisms behind ischemic post-conditioning. This study will pair clinical human data with molecular data. It is a novel theoretical concept in the field and the investigators believe that this methodology will be the basis for future research.

The investigators will utilize metabolomics as a tool to gain mechanistic insight into the potential mechanisms of action behind ischemic conditioning. Metabolomics is a burgeoning field of molecular biology that studies the metabolome, the catalogue of material and product of every biochemical reactions in the body occurring at that point in time. As such, the metabolome is ever changing and can reflect what the body is doing, not doing or responding to, and if so, by how much for each of the over 2,500 known human metabolites. Because there is such a large amount of data available by this technique, proper analysis requires the use of proprietary statistical software that can account for the effect of random chance in the data.

The particular innovation to this methodology compared to other studies to date is that we will pair biological as well as clinical data for analysis. This means that even if the investigators cannot find a difference in troponin levels between the treatment and control groups, the investigators will have some data on where to investigate next and be able to detect the biological response that remote post-ischemic conditioning induces. If this particular therapy does not develop any further, at least the investigators will know what appropriate mechanisms are at work and perhaps some of those could be targeted by pharmaceuticals in the future. Finally, if the investigators detect no differences at all, this will serve as an argument against the potential of ischemic post-conditioning in the NSTEMI population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 ≥ years old in the BIDMC ED
* Clinical suspicion of myocardial infarction
* ECG without pathognomonic ST-segment elevation
* At least one positive troponin-T (>0.10)

Exclusion Criteria:

* Inability to consent to enrollment
* Concurrent diagnosis of an emergent condition that may be antecedent to the NSTEMI
* Presentation to the ED greater than 24 hours after onset of NSTEMI symptoms
* Patients with a history of mastectomy or upper extremity arteriovenous fistula.
* Patients with active medication administration in both arms will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Changes in the Metabolomic Profile | Time: 0 minutes (baseline), 60 minutes, 2 hours, 3 hours, 24 hours, and 72 hrs.
  The change in metabolic profiles as compared to a subject's baseline readout will be analyzed using both, an "untargeted" and a "targeted" approach. A comparison of the these changes will be made between the interventional and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Shapiro, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
We may make the de-identified data available.

REFERENCES:
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction); American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Academic Emergency Medicine. ACC/AHA 2007 guidelines for the management of patients with unstable angina/non-ST-Elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction) developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. J Am Coll Cardiol. 2007 Aug 14;50(7):e1-e157. doi: 10.1016/j.jacc.2007.02.013. No abstract available. PMID 17692738
- [Background] Walsh M, Whitlock R, Garg AX, Legare JF, Duncan AE, Zimmerman R, Miller S, Fremes S, Kieser T, Karthikeyan G, Chan M, Ho A, Nasr V, Vincent J, Ali I, Lavi R, Sessler DI, Kramer R, Gardner J, Syed S, VanHelder T, Guyatt G, Rao-Melacini P, Thabane L, Devereaux PJ; Remote IMPACT Investigators. Effects of remote ischemic preconditioning in high-risk patients undergoing cardiac surgery (Remote IMPACT): a randomized controlled trial. CMAJ. 2016 Mar 15;188(5):329-336. doi: 10.1503/cmaj.150632. Epub 2015 Dec 14. PMID 26668200
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Background] Piot C, Croisille P, Staat P, Thibault H, Rioufol G, Mewton N, Elbelghiti R, Cung TT, Bonnefoy E, Angoulvant D, Macia C, Raczka F, Sportouch C, Gahide G, Finet G, Andre-Fouet X, Revel D, Kirkorian G, Monassier JP, Derumeaux G, Ovize M. Effect of cyclosporine on reperfusion injury in acute myocardial infarction. N Engl J Med. 2008 Jul 31;359(5):473-81. doi: 10.1056/NEJMoa071142. PMID 18669426
- [Background] Staat P, Rioufol G, Piot C, Cottin Y, Cung TT, L'Huillier I, Aupetit JF, Bonnefoy E, Finet G, Andre-Fouet X, Ovize M. Postconditioning the human heart. Circulation. 2005 Oct 4;112(14):2143-8. doi: 10.1161/CIRCULATIONAHA.105.558122. Epub 2005 Sep 26. PMID 16186417
- [Background] Vinten-Johansen J. Postconditioning: a mechanical maneuver that triggers biological and molecular cardioprotective responses to reperfusion. Heart Fail Rev. 2007 Dec;12(3-4):235-44. doi: 10.1007/s10741-007-9024-3. PMID 17520362
- [Background] Zhou Y, Fathali N, Lekic T, Ostrowski RP, Chen C, Martin RD, Tang J, Zhang JH. Remote limb ischemic postconditioning protects against neonatal hypoxic-ischemic brain injury in rat pups by the opioid receptor/Akt pathway. Stroke. 2011 Feb;42(2):439-44. doi: 10.1161/STROKEAHA.110.592162. Epub 2010 Dec 23. PMID 21183744
- [Background] Hausenloy DJ. Signalling pathways in ischaemic postconditioning. Thromb Haemost. 2009 Apr;101(4):626-34. PMID 19350104
- [Background] Mamas M, Dunn WB, Neyses L, Goodacre R. The role of metabolites and metabolomics in clinically applicable biomarkers of disease. Arch Toxicol. 2011 Jan;85(1):5-17. doi: 10.1007/s00204-010-0609-6. Epub 2010 Oct 16. PMID 20953584
- [Background] Montalescot G, Cayla G, Collet JP, Elhadad S, Beygui F, Le Breton H, Choussat R, Leclercq F, Silvain J, Duclos F, Aout M, Dubois-Rande JL, Barthelemy O, Ducrocq G, Bellemain-Appaix A, Payot L, Steg PG, Henry P, Spaulding C, Vicaut E; ABOARD Investigators. Immediate vs delayed intervention for acute coronary syndromes: a randomized clinical trial. JAMA. 2009 Sep 2;302(9):947-54. doi: 10.1001/jama.2009.1267. PMID 19724041
- [Background] Alcalai R, Planer D, Culhaoglu A, Osman A, Pollak A, Lotan C. Acute coronary syndrome vs nonspecific troponin elevation: clinical predictors and survival analysis. Arch Intern Med. 2007 Feb 12;167(3):276-81. doi: 10.1001/archinte.167.3.276. PMID 17296884